CLINICAL TRIAL: NCT05340296
Title: Network Health Intervention for Adolescents Leaving Acute Psychiatric Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funds remained for additional recruitment
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Ian Cero, Senior Instructor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006651; 2KL2TR001999-05 (NIH); https://osf.io/8pd54/ (Other: Open Science Foundation)
Record Dates: First submitted 2022-03-03; First posted 2022-04-22 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Suicide, Attempted
Keywords: suicide; suicide attempt; suicide ideation; adolescent; social network
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Intervention Model Description: All subjects will receive Acute Youth Connect plus treatment as usual.
Masking Description: There is only one arm. No masking will be attempted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute Youth Connect + TAU (Experimental): Subjects will receive 12 weeks of post-discharge Acute Youth Connect intervention, in addition to regular post-discharge treatment as usual.
  Interventions: Behavioral: Acute Youth Connect

INTERVENTIONS:
Behavioral: Acute Youth Connect — This intervention is being piloted will be revised with feedback from the first 5-10 patients who complete it. At the time of registration, the protocol is as follows: Roughly one week prior to discharge, the patient and a parent/caregiver will together nominate 3-4 trusted adults in the patient's life to serve as their post-discharge support team. Consenting nominees will then attend a 45-90 minute training on how to provide social support to the patient. Each adult support will also receive weekly (3-15 minute) check in calls from study staff to monitor progress and concerns. Each patient will also attend 3 interactive sessions with a study interventionist, and will be encouraged to bring an adult from their support team. These sessions will be evenly spaced throughout the post-discharge intervention period. Adolescents will receive weekly reflection-prompting text messages to practice skills taught in the interactive sessions.

SUMMARY:
The purpose of this pilot study is to refine and then assess the feasibility, acceptability, and target engagement of Acute Youth Connect - a network health intervention for adolescents leaving acute psychiatric care with suicide-related concerns.

DETAILED DESCRIPTION:
This pilot study includes only one arm of subjects, all of whom will receive Acute Youth Connect, in addition to treatment as usual. The Acute Youth Connect treatment protocol lasts for 12 weeks following discharge, for a total intervention period of roughly 13 weeks including pre-discharge consent and nomination of supports. Patients will be assessed at baseline, mid-intervention, immediately post-intervention, and 12 weeks following the scheduled intervention completion.

Feedback from the first 5-10 patients will be used to modify the treatment protocol to improve patient acceptability. All remaining patients will receive this refined treatment protocol.

At the time of registration, the Acute Youth Connect treatment protocol is as follows. Adolescents in acute psychiatric care (partial hospitalization) will be screened for eligibility approximately one week before discharge. After patient assent and parental consent are received, the patient and a parent/caregiver will together nominate 3-4 trusted adults in the patient's life to serve as a post-discharge support team. The nominees will then be contacted, consented, and receive a 45-90 minute training on how to provide social support to the patient. Each adult support will also receive weekly (3-15 minute) check in calls from study staff to monitor progress and resolve any concerns related to the patient's progress. In addition, each patient will attend 3 interactive sessions with a study interventionist, and will be encouraged to bring an adult from their support team to participate as well. These sessions will be evenly spaced throughout the post-discharge intervention period. Adolescents will receive weekly reflection-prompting text messages to practice skills taught in the interactive sessions.

ELIGIBILITY:
Youth subjects will be included if:

* Youth subject is being discharged from the Child and Adolescent Partial Hospital Service (CAPHS) in the URMC Department of Psychiatry.
* Youth subject endorses past year suicide attempt OR past year suicidal ideation at time of partial hospitalization, as assessed on standardized intake questionnaire used by CAPHS.
* Youth subject has a cellular phone, with an active service plan, that is capable of sending and receiving standard SMS text messages.
* Youth subject is aged 12 - 18 at time of enrollment.

Youth subjects will be excluded if:

* Youth subject has medical or psychiatric comorbidities that impair ability to assent (e.g., active psychotic or manic episode, cognitive impairment).
* Youth subject patient or guardian does not speak fluent English, as meeting translation costs is not possible in this study.
* Youth subject is unable to name at least 2 trusted adults (at least 1 of which is not a parent or caregiver) they would like to serve on their support team.
* Youth is unable or unwilling to share their suicide-related safety plan

Parent / legal guardian subjects will be included if:

- Adult subject is at least 21 years of age.

Adult support team subjects will be included if:

* Adult subject is nominated by a youth subject to serve on their adult support team
* Adult subject is approved by youth subject's parent or legal guardian
* Adult subject has a cellular phone, with an active service plan, that is capable of sending and receiving standard SMS text messages.
* Adult subject is at least 21 years of age.

Adult support team subjects will be excluded if:

* Adult subject has medical or psychiatric comorbidities that impair ability to consent (e.g., active psychotic or manic episode, cognitive impairment).
* Adult subject does not speak fluent English, as meeting translation costs is not possible in this study.
* Adult reports being unable to be in contact with youth at least once per week, for the 12 weeks of the intervention

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Number of youth who complete the intervention | Interactive sessions by the end of the 12-week intervention.
  Youth subjects who complete all three interactive sessions will be marked as "treatment completers."
Text message responses | A text message must be responded to before the next text message prompt is sent (roughly one week).
  Text message prompts will be marked as "responded to" when a recipient produces at least one reply.
Adult support team treatment completion | Psychoeducation sessions must be completed before week 4 after youth's discharge. Check-in calls must be completed in seperatecalendar weeks, all before the end of the 12-week intervention.
  Adult support team members who complete their initial psychoeducation training session and complete 75% of their check-in phone calls will be marked as "treatment completers".

SECONDARY OUTCOMES:
Change in weekly contact to supportive adults in their lives | Baseline to post-treatment, approximately 3 months
  Youth subjects will report a change in the average weekly contact with the members of their adult support team, compared to reported baseline contact.
Change in weekly contact to supportive adults in their lives | Baseline to 3 months post-treatment, approximately 6 months
  Youth subjects will report a change in the average weekly contact with the members of their adult support team, compared to reported baseline contact.
Utilization of intervention content | Baseline to post-treatment, approximately 3 months
  Rate of adolescents reporting using at least two of the three Acute Youth Connect cores (connection, balance, purpose) weekly or more.
Utilization of intervention content | Baseline to 3 months post-treatment, approximately 6 months
  Rate of adolescents reporting using at least two of the three Acute Youth Connect cores (connection, balance, purpose) weekly or more.

OTHER OUTCOMES:
Change in perceived social connectedness | Baseline to post-treatment, approximately 3 months
  Interpersonal Needs Questionnaire - Belongingness subscale. Total scores range from 0-54, higher scores indicate more social distress. We predict a change in distress.
Change in perceived social connectedness | Baseline to 3 months post-treatment, approximately 6 months
  Interpersonal Needs Questionnaire - Belongingness subscale. Total scores range from 0-54, higher scores indicate more social distress. We predict a change in distress.
Change in feelings of meaning | Baseline to post-treatment, approximately 3 months
  Claremont Purpose Scale - Personal Meaning subscale. Total scores range from 0-16 for each subscale scale. Higher scores indicate more feelings of meaning and purpose. We predict a change in scores on each subscale.
Change in feelings of meaning | Baseline to 3 months post-treatment, approximately 6 months
  Claremont Purpose Scale - Personal Meaning subscale. Total scores range from 0-16 for each subscale scale. Higher scores indicate more feelings of meaning and purpose. We predict a change in scores on each subscale.
Change in feelings of purpose | Baseline to post-treatment, approximately 3 months
  Claremont Purpose Scale - Goal-directedness subscale. Total scores range from 0-16 for each subscale scale. Higher scores indicate more feelings of meaning and purpose. We predict a change in scores on each subscale.
Change in feelings of purpose | Baseline to 3 months post-treatment, approximately 6 months
  Claremont Purpose Scale - Goal-directedness subscale. Total scores range from 0-16 for each subscale scale. Higher scores indicate more feelings of meaning and purpose. We predict a change in scores on each subscale.
Changes in interpersonal emotion regulation | Baseline to post-treatment, approximately 3 months
  Interpersonal Emotion Regulation Questionnaire - Social Modeling Subscale (scores range from 5-25, higher scores indicate improved functioning). We predict a change in scores.
Changes in interpersonal emotion regulation | Baseline to 3 months post-treatment, approximately 6 months
  Interpersonal Emotion Regulation Questionnaire - Social Modeling Subscale (scores range from 5-25, higher scores indicate improved functioning). We predict a change in scores.
Changes in access to emotion regulation strategies | Baseline to post-treatment, approximately 3 months
  Difficulties in Emotion Regulation Scale - Regulation Strategies Subscale (scores range from 3-15, higher scores indicate greater dysfunction). We predict a change in scores.
Changes in access to emotion regulation strategies | Baseline to 3 months post-treatment, approximately 6 months
  Difficulties in Emotion Regulation Scale - Regulation Strategies Subscale (scores range from 3-15, higher scores indicate greater dysfunction). We predict a change in scores.
Changes in engagement with healthy activities | Baseline to post-treatment, approximately 3 months
  Behavioral Activation for Depression - Short form - Activation Subscale. Scores range from 5-35, with higher scores indicating greater function. We predict a change in function.
Changes in engagement with healthy activities | Baseline to 3 months post-treatment, approximately 6 months
  Behavioral Activation for Depression - Short form - Activation Subscale. Scores range from 5-35, with higher scores indicating greater function. We predict a change in function.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Cero, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD with other researchers.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT05340296/Prot_SAP_ICF_000.pdf